CLINICAL TRIAL: NCT00664313
Title: TBTC Study 30: A Phase I/II Pilot Study for Evaluation of Low Dose, Once Daily, Linezolid Plus Optimized Background Therapy (OBT) Versus Placebo Plus OBT for the Treatment of Multi-drug Resistant Tuberculosis
Brief Title: TBTC Study 30: Safety and Tolerability of Low Dose Linezolid in MDR TB
Acronym: LiMiT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of KwaZulu (Other); Columbia University (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDC-NCHHSTP-5356; NCT00691392 (obsolete NCT alias)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Multi-drug Resistant Tuberculosis; Extensively Drug Resistant Tuberculosis
Keywords: Linezolid; Zyvox; Peripheral Neuropathy; Optic Neuropathy; Anemia; Thrombocytopenia
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis; Peripheral Nervous System Diseases; Optic Nerve Diseases; Anemia; Thrombocytopenia | interventions — Linezolid; stearic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linezolid (Experimental): Linezolid 600 mg po QD
  Interventions: Drug: Linezolid
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linezolid — 600 mg po daily for 112 doses (16 weeks)
  Other Names: Zyvox
  Arms: Linezolid
Drug: Placebo — Placebo given daily for 112 doses (16 weeks)
  Other Names: PH-102 Avicel (96%), Explotab sodium starch glycolate (3%), and Magnesium stearate (1%)
  Arms: Placebo

SUMMARY:
The antibiotic linezolid when given for the treatment of multi-drug resistant tuberculosis is safe and tolerated at a low dose (600 mg daily) for a limited duration (16 weeks)

ELIGIBILITY:
Inclusion Criteria

1. Pulmonary tuberculosis with or without extrapulmonary TB with a M. tuberculosis isolate that is confirmed to be resistant to at least rifampin and isoniazid (without regard to prior treatment for TB).
2. A documented positive sputum culture result for M. tuberculosis from a sputum obtained in the four months prior to enrollment.
3. Willingness to have HIV testing performed, if HIV serostatus is not known or if the last documented negative HIV test was more than 6 months prior to enrollment.
4. Residence within the Durban Functional Region (Durban Metropolitan Area) or Tugela Ferry, Msinga District, KZN, RSA.
5. Age ≥ 18 years.
6. Karnofsky score of > 50 (see section 18.1)
7. Willingness by the patient to attend scheduled follow-up visits and undergo study assessments.
8. Women with child-bearing potential must agree to practice an adequate method of birth control or to abstain from heterosexual intercourse during study therapy. (Standard birth control measures are provided free of charge by public health institutions)
9. Laboratory parameters done within 14 days prior to screening:

   1. Serum creatinine level < 2 times upper limit of normal
   2. Hemoglobin level ≥ 9.0 g/dL
   3. Platelet count of ≥ 80,000/mm3
   4. Absolute neutrophil count (ANC) > 1000/ mm3
   5. Negative pregnancy test (for women of childbearing potential)
10. Able to provide informed consent or legally authorized representative able to do so if decisionally impaired.

Exclusion Criteria

1. Currently breast-feeding or pregnant.
2. Known allergy or intolerance to linezolid.
3. Planned therapy during the intensive phase of tuberculosis treatment using drugs having unacceptable interactions with linezolid, including dopamine, selective serotonin uptake inhibitors (citalopram, fluoxetine, fluvoxamine, paroxetine, and sertraline), amitriptyline, bupropion, mirtazepine, levodopa, carbidopa, sinemet, or herbal medications.
4. Significant peripheral neuropathy as evidenced by < 5 seconds of vibratory sense to a 128 Hz tuning fork on either big toe
5. Pain, aching or burning of the feet that interfere with walking or sleep.
6. In the judgment of the physician the patient is not expected to survive for more than 4 weeks.
7. Anticipated surgical intervention for the treatment of pulmonary tuberculosis
8. Visual acuity of 20/200 (6/60 meters) best corrected vision or less.
9. Poor color vision as evidenced by incorrect answers on > four of 12 screening Ishihara plates
10. Participation in another drug trial.
11. The patient has received second line TB drugs for > 7 days immediately prior to enrollment (note: use of first line drugs such as INH, Rifampin, PZA, or ethambutol for > 7 days immediately prior to enrollment is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Cumulative rate of serious adverse events - SAEs (measured as the number of SAEs per person days) during the period of study therapy and the four weeks of post-study therapy follow-up. | the period of study therapy (generally 16 weeks) plus the four weeks of post-study therapy follow-up.
Proportion of patients in each arm who complete 80% of the proposed regimen (90 doses) within 18 weeks of treatment initiation. | within 18 weeks of treatment initiation

SECONDARY OUTCOMES:
The number of days required to convert to culture negative status in sputum of those in each treatment arm on solid and liquid media, respectively. | first 16 weeks of study therapy
The proportion of culture-negative patients during the first 16 weeks of therapy (at two week intervals) of linezolid with OBT vs. that of OBT with placebo on solid and liquid media, respectively | first 16 weeks of study therapy
Time to detection of M. tuberculosis on MGIT for each positive culture for sputum specimens collected every 2 weeks during the first 16 weeks of therapy | First 16 weeks of study therapy
The occurrence of treatment failure in the first 12 month following initiation of study therapy | first 12 months
Changes from baseline in assessments for peripheral neuropathy | First 12 months
Changes from baselines in Snellen or Jaeger visual acuity test and Ishihara color plate test results to assess for optic neuropathy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Saukkonen, MD, Principal Investigator — Boston University; Waffa El-Sadr, MD, Principal Investigator — Columbia University; Nesri Padayachin, MBChB, Principal Investigator — University of Kwa-Zulu Natal
Locations (1):
- King George V Hospital, Durban, South Africa

REFERENCES:
- [Derived] Padayatchi N, Mac Kenzie WR, Hirsch-Moverman Y, Feng PJ, Villarino E, Saukkonen J, Heilig CM, Weiner M, El-Sadr WM. Lessons from a randomised clinical trial for multidrug-resistant tuberculosis. Int J Tuberc Lung Dis. 2012 Dec;16(12):1582-7. doi: 10.5588/ijtld.12.0315. PMID 23131255